CLINICAL TRIAL: NCT00641446
Title: Rates of Seroconversion Following Varicella Vaccination of Asthmatic Children Between the Ages of One and Eight Years Treated With Pulmicort Respules® Versus Non-Steroidal Conventional Asthma Therapy
Brief Title: Varicella Vaccination With Pulmicort
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Lars-Göran Carlsson
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SD-004-0758; D5257C00758
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: Children; Asthma; Varivax; varicella; Pulmicort; budesonide
MeSH Terms: conditions — Asthma; Chickenpox | interventions — Budesonide; Chickenpox Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pulmicort
  Interventions: Drug: budesonide
- 2 (Active Comparator): Varivax
  Interventions: Drug: varicella zoster virus

INTERVENTIONS:
Drug: budesonide
  Other Names: Pulmicort
  Arms: 1
Drug: varicella zoster virus
  Other Names: Varivax
  Arms: 2

SUMMARY:
A study to determine whether treatment with Pulmicort in children has any effect on the varicella vaccine

ELIGIBILITY:
Inclusion Criteria:

* Children between the age of 10 months and 8 years,
* have asthma or shown recent signs suggesting asthma,
* have a parent or guardian willing to comply with study requirements

Exclusion Criteria:

* Varicella zoster immune globulin (VZIG) within 5 months prior to immunization,
* Previous varicella immunization,
* an immunization or allergy immunotherapy 4 weeks prior to immunization,
* Severe asthma,
* have another persistent lung disease,
* have a planned hospitalization for the duration of study

Ages: 10 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2001-10; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Seroconversion level | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Bertill Andersson, Study Director — AstraZeneca employee